CLINICAL TRIAL: NCT05566431
Title: Pediatric Severe Traumatic Brain Injury in Latin America - A Randomized Trial Comparing Two Management Protocols
Brief Title: Benchmark Evidence Led by Latin America: Trial of Intracranial Pressure - Pediatrics
Acronym: BELA TRIPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Randall M. Chesnut, Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00013122; 1R01HD106273-01 (NIH)
Record Dates: First submitted 2022-06-10; First posted 2022-10-04 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Severe Traumatic Brain Injury
Keywords: sTBI; ICP monitoring; randomized controlled trial; TBI management; Latin America; pediatric; Phase III
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: In a Phase III multicenter, parallel-group, randomized superiority trial in 428 children with sTBI from 7 Latin American pediatric trauma centers, the objective is to test the efficacy of the treatment protocol from the Guidelines based on ICP monitoring among children with sTBI in improving global outcome measured by Pediatric Quality of Life Inventory (PedsQL) 6 mos after injury compared to treatment based on a non-invasive imaging & clinical examination (CREVICE) protocol specifically modified for a pediatric population.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will not go into the ICU when a study participant is being treated, unmasked study staff will not inform the outcome assessor which protocol was used for a participant. and outcome assessors will remind participant's parents to refrain for telling them which treatment protocol was used for the participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ICP monitoring based Protocol (Active Comparator): Arm one will use a consensus-developed management protocol for paediatric severe traumatic brain injury based on recommendations from the Brain Trauma Foundation Guidelines, which uses invasive intracranial pressure monitoring
  Interventions: Other: ICP
- No ICP Monitoring Protocol CREVICE (Active Comparator): Arm two will use the Consensus-Revised Imaging and Clinical Examination (CREVICE) management protocol for paediatric severe traumatic brain injury based on imaging and clinical examination in the absence of invasive intracranial pressure monitoring
  Interventions: Other: CREVICE

INTERVENTIONS:
Other: ICP — The intervention is a management protocol that includes ICP monitoring for children with severe traumatic brain injury
  Other Names: Intracranial-pressure-monitoring-based management protocol
  Arms: ICP monitoring based Protocol
Other: CREVICE — The intervention is a management protocol that is based on imaging and clinical examinations without ICP monitoring for children with severe traumatic brain injury
  Other Names: Imaging-and-clinical-examination-based management protocol
  Arms: No ICP Monitoring Protocol CREVICE

SUMMARY:
Narrative:

Worldwide, traumatic brain injury (TBI) is a leading cause of death and disability among children and adolescents. The Investigators aim to test whether pediatric TBI treatment guided by invasive intracranial pressure monitoring produces better patient outcomes than care guided by a protocol without invasive monitoring. Study findings will inform clinical practice in treating pediatric severe TBI globally. Focused didactic and experience-based learning opportunities will increase the research capacity of pediatric intensivists in Latin America.

DETAILED DESCRIPTION:
Abstract:

Children who survive severe traumatic brain injury (sTBI) live with profound impairments that alter their development and future possibilities. Worldwide, TBI is the leading cause of death and disability for children/ adolescents with the US annual incidence 6 times greater than MS, HIV/AIDS, spinal cord injury, and breast cancer combined.

Our primary focus for scientific investigation is to conduct a high quality randomized controlled trial addressing a critical TBI management question: Does using a protocol with information from intracranial pressure (ICP) monitoring to direct treatment of children with sTBI improve outcomes vs an aggressive management protocol based on imaging and clinical examination alone? This follows on our adult ICP study which found no outcome differences and has occasioned re-thinking of treatment guidelines for sTBI patients >13. A separate study is essential because children are not simply small adults and some treatment approaches carry age-related additional risks. Thus, study findings will inform US and global clinical practice.

This trial will be conducted in 8 Latin American pediatric ICUs where infrastructures and practice patterns are optimal for strong internal validity and resources represent trauma care in the developing world. The successful adolescent/adult BEST TRIP trial, which collected high-quality data in similar environments (cited > 900 times) underscores the feasibility of this approach.

Specific Aim: In a Phase III randomized superiority trial in 428 children with sTBI from 8 Latin American pediatric trauma centers, test the effect on outcomes of management of sTBI guided by a protocol using information from ICP monitors vs. management using a protocol that uses imaging and clinical exams to guide treatment.

Hypothesis #1: Children with severe TBI whose acute care treatment is managed using a protocol based on data from ICP monitoring will have significantly lower mortality and better quality of life and global outcome at 6 months post-trauma than those whose treatment is managed with a protocol based on imaging and clinical exam. The primary measure of functional recovery is the PedsQL at 6 months. A secondary measure is GOSE-Peds.

Hypothesis #2: Incorporating ICP monitoring into sTBI patient care will minimize secondary complications, decrease length of stay in ICU and decrease brain-specific treatments.

Specific Aim: The Investigators will train personnel in centers new to research how to conduct high-quality scientific studies, and will extend the training for the personnel with whom the Investigators have been working, solidifying previous capacity-building efforts, and initiating new efforts.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form by the parent(s) or guardian(s)
2. Non-penetrating TBI
3. Admission to study hospital within 24 hours of injury
4. Total GCS score ≤ 8 on admission or within first 48 hours after injury (measured using pediatric GCS 1 for children < 2 years old and standard GCS for older children)
5. Age 1 through 12 years
6. Able to randomize:

   * Within 24 hours of injury (for patients with GCS ≤ 8 on admission) OR
   * Within 24 hours of deterioration (for patients deteriorating to GCS ≤ 8 within 48 hours of injury)

Exclusion Criteria:

1. Motor GCS score of 6
2. GCS of 3 with bilaterally fixed and dilated pupils
3. Injury thought to be intentionally inflicted by a family member or caregiver.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 428 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Pediatric Quality of Life Inventory (PedsQL) | 6 months after injury
  PedsQL is a generic, health-related quality of life instrument developed to measure the core dimensions of physical, cognitive, mental, social health, and role (school) function. Minimum and maximum values: 0-100. Higher scores have better outcomes.

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory (PedsQL) | 3 months after injury
  PedsQL is a generic, health-related quality of life instrument developed to measure the core dimensions of physical, cognitive, mental, social health, and role (school) function. Minimum and maximum values: 0 - 100. Higher the score means a better outcome.
Glasgow Outcome Scale - Extended (GOS-E) Pediatric | 3 and 6 months after injury
  GOS-E is the most common measure of functional outcome in adult TBI trials. Its pediatric version is the primary outcome in the NINDS-funded ADAPT study. Minimum and maximum values: 1-8. Higher score has worse outcomes.
Mortality | 3 and 6 months
  Percent of participants who have died by the assessment time.
Brain-specific interventions | 1 month average
  Total number of individual interventions directed at treating measured or suspected intracranial hypertension (i.e., brain-specific treatment) per hour summed over the duration of brain-specific treatment in ICU. Time Frame for brain-specific treatments is through acute hospitalization, an average of one (1) month and for GOS-E Peds is conducted 3 and 6 months after injury.
ICU length of stay | 1 month average
  ICU length of stay related to TBI management is through acute hospitalization and for an average of one (1) month.

CONTACTS AND LOCATIONS:
Overall Officials: Randall Chesnut, MD, Principal Investigator — University of Washington
Locations (11):
- University of Washington, Harborview Medical Center, Seattle, Washington, United States
- Colombia (2):
  - Fundación Hospital de la Misericordia, Bogotá
  - Hospital Fundacion Amigos de la Salud, Montería
- Hospital de Niños Benjamín Bloom, San Salvador, El Salvador
- Guatemala (3):
  - Hospital Regional de Esquintla, Escuintla
  - Hospital General San Juan de Dios, Guatemala City
  - Hospital Regional de Occidente San Juan de Dios, Quetzaltenango
- Hospital Escuela, Tegucigalpa, Honduras
- Peru (3):
  - Hospital de Emergencias Pediátricas, Lima
  - Hospital Edgardo Rebagliati Martins, Lima
  - Instituto Nacional de Salud del Niño - San Borja, Lima

IPD SHARING:
Plan to Share IPD: Yes
When the study is completed, access to study data may be provided through the UW Data Repository for future analyses about brain injury, its treatment, and outcomes or other scientifically appropriate questions. A de-identified dataset will be provided to successful candidates for the specified use.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available 1 year after the primary study results are published.
Access Criteria: Researchers will complete a data use agreement that includes the questions to be answered with the data.

REFERENCES:
- [Derived] Chesnut R, Temkin N, Pridgeon J, Sulzbacher S, Lujan S, Videtta W, Moya-Barquin L, Chaddock K, Bonow RH, Petroni G, Guadagnoli N, Hendrickson P, Ramirez Cortez G, Carreazo NY, Vargas Aymituma A, Anchante D, Caqui P, Ramirez A, Munaico Abanto M, Ortiz Chicchon M, Cenzano Ramos J, Castro Darce MDC, Sierra Morales R, Brol Lopez P, Menendez W, Posadas Gutierrez S, Kevin V, Mazariegos A, de Leon E, Rodas Barrios RE, Rodriguez S, Flores S, Alvarado O, Guzman Flores LJ, Moisa Martinez M, Gonzalez P. Development of a Randomized Trial Comparing ICP-Monitor-Based Management of Severe Pediatric Traumatic Brain Injury to Management Based on Imaging and Clinical Examination Without ICP Monitoring-Research Algorithms. Neurosurgery. 2024 Jan 1;94(1):72-79. doi: 10.1227/neu.0000000000002760. Epub 2023 Nov 13. PMID 37955439
- [Derived] Chesnut R, Temkin N, Pridgeon J, Sulzbacher S, Lujan S, Videtta W, Moya-Barquin L, Chaddock K, Bonow R, Petroni G, Guadagnoli N, Hendrickson P, Ramirez Cortez G, Carreazo NY, Vargas Aymituma A, Anchante D, Caqui P, Ramirez A, Munaico Abanto M, Ortiz Chicchon M, Cenzano Ramos J, Mazate-Mazariegos A, Castro Darce MDC, Sierra Morales R, Brol Lopez P, Menendez W, Posadas Gutierrez S, Kevin V, Mazariegos A, de Leon E, Rodas Barrios RE, Rodriguez S, Flores S, Alvarado O, Guzman Flores LJ, Moisa Martinez M, Gonzalez P. Development of a Randomized Trial Comparing ICP-Monitor-Based Management of Severe Pediatric Traumatic Brain Injury to Management Based on Imaging and Clinical Examination Without ICP Monitoring-Study Protocol. Neurosurgery. 2024 Jan 1;94(1):65-71. doi: 10.1227/neu.0000000000002582. Epub 2023 Jul 6. PMID 37409817